CLINICAL TRIAL: NCT06940791
Title: Tirabrutinib Maintenance Versus Placebo in Patients With Primary Central Nervous System Lymphoma in Complete Remission: a Randomized Phase II Study (JCOG2104)
Brief Title: Tirabrutinib Maintenance Versus Placebo in Patients With Primary CNS Lymphoma in Complete Remission (JCOG2104)
Acronym: TIMELY-pII
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyorin University (Other)
Collaborators: National Cancer Center, Japan (Other Government); Ono Pharmaceutical Co. Ltd (Industry); Japan Clinical Oncology Group (Other)
Responsible Party: Principal Investigator, Motoo Nagane, Professor, Department of Neurosurgery, Kyorin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JCOG2104
Record Dates: First submitted 2025-04-04; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — tirabrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard arm (Placebo Comparator): Observation with placebo
  Interventions: Drug: Placebo
- Experimental arm (Experimental): Tirabrutinib maintenance therapy
  Interventions: Drug: Tirabrutinib

INTERVENTIONS:
Drug: Tirabrutinib — Tirabrutinib (480 mg) taken orally daily at fasting condition
  Arms: Experimental arm
Drug: Placebo — Placebo taken orally daily at fasting condition
  Arms: Standard arm

SUMMARY:
A double-blind, randomized phase II comparative trial will evaluate the superiority of the investigational treatment (tirabrutinib maintenance therapy) over standard care (observation with placebo) in terms of progression-free survival in patients with newly diagnosed primary central nervous system lymphoma (PCNSL) who have achieved complete response (CR or CRu) following induction therapy with high-dose methotrexate (HD-MTX)-based chemotherapy and have not undergone consolidative whole-brain irradiation.

Participants will:

Take protocol drug tirabrutinib or a placebo every day until disease progression or experience of unacceptable toxicity.

Visit the clinic once every 4 weeks for checkups and tests, as well as protocol drug prescription.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological diagnosis of B cell lymphoma.
2. Newly-diagnosed PCNSL confined to the cerebrum, cerebellum and brainstem. Patients with or without interocular lymphoma are eligible.
3. Negative cerebrospinal fluid (CSF) cytology, or no evidence of leptomeningeal lymphomatosis in contrast-enhanced magnetic resonance imaging (MRI) of the brain and the whole spinal cord.
4. No evidence of systemic lymphoma before induction chemotherapy, confirmed by contrast-enhanced CT including the neck, chest, abdomen, pelvic cavity and groin, or whole-body positron-emission tomography (PET) and CT.
5. Patients with a single lesion, or multiple lesions, are eligible.
6. Patients 18 years old or older at the time of registration.
7. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0, 1, 2.
8. Have completed either of the following methotrexate (MTX)-based chemotherapy i) R-MPV (rituximab, MTX, procarbazine and vincristine) ii) MPV (MTX, procarbazine and vincristine) iii) R-MP (rituximab, MTX and procarbazine) iv) MP (MTX and procarbazine) v) R-M (rituximab and MTX) vi) MTX monotherapy
9. Complete response (CR) or complete response unconfirmed (CRu) based on the International PCNSL Collaborative Group (IPCG) criteria.
10. Within 60 days from the last dose of induction or consolidation chemotherapy.
11. No treatment history of radiotherapy for PCNSL.
12. Refused to receive consolidation radiotherapy.
13. No treatment history of chemotherapy or radiotherapy, except for stereotactic radiosurgery (SRS) or stereotactic radiotherapy (SRT) for non-cancer diseases (such as arteriovenous malformations).
14. Adequate organ function. i) Neutrophil count >=1,000/mm3 ii) Hemoglobin >= 8.0 g/dl iii) Platelet count >= 75,000/mm3 iv) AST <=120 U/L v) ALT <= 120 U/L vi) Total Bilirubin <= 2.25 mg/dl vii) Creatinine <= 1.5 mg/dL
15. Written informed consent.

Exclusion Criteria:

1. Synchronous or metachronous malignancies.
2. Infections requiring systemic treatment at the time of registration.
3. Body temperature >=38 degree celsius at the time of registration.
4. Serious lung disorders, such as interstitial pneumonia, obstructive lung disease, hypersensitive pneumonitis, symptomatic bronchospasm) at the time of registration.
5. History or presence of aspergillus pneumonitis or pneumocystis pneumonia.
6. History of serious drug allergy or serious anaphylaxis.
7. Heart failure (>= III in New York Heart Association functional classification), unstable angina pectoris, or history of myocardial infarction within the preceding 180 days prior to registration.
8. Treated by anticoagulants at the time of registration.
9. Treated by antiplatelets at the time of registration.
10. Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP).
11. Immune deficiency, such as acquired immunodeficiency syndrome (AIDS), X-linked agammaglobulinemia, chronic granulomatous disease, Wiskott-Aldrich syndrome, or any other iatrogenic immunosuppressive conditions.
12. Post organ transplant immunosuppression.
13. Prednisone use of >10 mg/day for condition other than intracranial tumor, or regular use of immunosuppressants.
14. Uncontrolled diabetes mellitus.
15. Treated either by CYP3A4 inhibitors, CYP3A4 inducers, or P-gp inducers within 14 days prior to registration.
16. Gadolinium allergy.
17. Positive HIV antibody.
18. Positive HBs antigen.
19. Positive HBs antibody or HBc antibody, and HBV-DNA positive.
20. Positive HCV antibody.
21. Unable to take oral medicine,
22. Females during pregnancy, or within 28 days postpartum, or during lactation. Males who wish childbearing of his partner.
23. Prior history of treatment by BTK inhibitors.
24. Severe psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) based on independent review committee (IRC) assessment | From the date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 78 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) determined by investigator | From the date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 78 months
Overall survival (OS) | From the date of registration until the date of death from any cause, assessed up to 78 months
PFS/OS in the maintenance per protocol group | PFS: From the date of registration until the date of first progression or date of death from any cause, whichever came first, assessed up to 78 months. OS: From the date of registration until the date of death from any cause, assessed up to 78 months.
PFS/OS by the induction therapy regimen with or without consolidation therapy | PFS: From the date of registration until the date of first progression or date of death from any cause, whichever came first, assessed up to 78 months. OS: From the date of registration until the date of death from any cause, assessed up to 78 months.
Incidence rate of adverse events | During the intervention up to 78 months, or for those who discontinued the intervention, assessed until 30 days after the last date of intervention or the date of initiation of post-study therapy, whichever came first, assessed up to 78 months.
  The proportion of patients who experienced each adverse event
Proportion of patients without neurological cognitive function (NCF) deterioration | Among patients eligible for NCF assessment, the proportion without deterioration in each assessment item at the following time points: pre-treatment baseline (after registration but before initiation of the study treatment), 48 weeks, 2 years, and 3 year
Proportion of patients without deterioration in health-related QOL | Among patients eligible for HR-QOL assessment, the proportion without deterioration at the following time points: pre-treatment baseline (after registration but before initiation of the study treatment), 48 weeks, 2 years, and 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kyorin University Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided